CLINICAL TRIAL: NCT01457976
Title: A Survey on Attitudes on Personal Responsibility and the Use of Financial Incentives for Health Promotion
Brief Title: A Survey on Attitudes on Financial Incentives
Status: Withdrawn | Type: Observational
Why Stopped: protocol never approved by local IRB
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 814399
Record Dates: First submitted 2011-09-21; First posted 2011-10-24 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Colon Cancer
Keywords: cancer; obesity; personal responsibility
MeSH Terms: conditions — Obesity; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Members of the US public, non-probability sample
- Members of the German public, non-probability sample
- Members of the US public, probability sample

SUMMARY:
The study concerns a survey of attitudes of the public on issues around personal responsibility for health and the use of financial incentives to promote health in the U.S. and Germany. All data are gathered anonymously through online platforms. Two separate professional panel providers are used for access to members of the public. All participants are people who have voluntarily joined a survey panel in the past through an informed consent process and currently serve as panel members.

ELIGIBILITY:
Inclusion Criteria:

* none other than age

Exclusion Criteria:

* none other than age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult American and Germans
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Survey respondents are presented with scenarios that seek to elicit views and attitudes on the concepts of personal responsibility, and the acceptability of financial incentives. The analysis will present these views and attitudes in aggregate form. | 2 weeks
  Attitudes are measured using 5 point Likert scales, indicating the extent of agreement or disagreement with particular scenarios or questions. Other forms of multiple choice options are also used, in which respondents express their preferences by selecting one option over others. At the end of the surveys, an open text box is provided for general comments.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, Ph.D, M.D., Principal Investigator — School of Medicine, University of Pennsylvania
Locations (1):
- Online survey, Philadelphia, Pennsylvania, United States